CLINICAL TRIAL: NCT00157261
Title: A Prospective, Randomised, Double-blind, Placebo-controlled, International, Multicentre, Parallel-group Comparison Trial Evaluating the Efficacy and Safety of Tenecteplase During Cardiopulmonary Resuscitation as Compared With Standard Treatment in Patients Suffering From Out-of-hospital Cardiac Arrest of Presumed Cardiac Origin Thrombolysis in Cardiac Arrest (TROICA) Trial
Brief Title: Thrombolysis Using Tenecteplase (Metalyse®) in Cardiac Arrest - The TROICA Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1123.18
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Heart Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Tenecteplase

INTERVENTIONS:
Drug: tenecteplase

SUMMARY:
The general aim of this study is to compare the efficacy and safety of tenecteplase to standard treatment during cardiopulmonary resuscitation in patients suffering from out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
The trial is a prospective, international, multi-centre, randomised (1:1), double-blind, parallel group comparison conducted for investigating the efficacy and safety of tenecteplase and placebo in patients with cardiac arrest of presumed cardiac origin.

Approximately 1300 patients (two groups of 650 patients; tenecteplase or matching placebo) suffering from witnessed (by eye or ear) out-of-hospital cardiac arrest of presumed cardiac origin, who are treated with ALS-CPR will be randomised at approximately 40 study centres. Randomisation is done immediately after insertion of an IV line is established. Study drug application, as a single IV bolus over 5-10 seconds, should be done immediately after the first vasopressor application during the ALS-CPR procedure.

PCI facilities will be required at all participating sites, i.e. hospitals receiving patients.

Study Hypothesis:

The primary aim of the trial is to demonstrate superiority in the intent-to-treat analysis of tenecteplase over placebo with regard to primary endpoint as the incidence of 30-day survival (30daysurv).

Comparison(s):

Group A (experimental; fibrinolytic treatment) Tenecteplase, as a single IV bolus over 5-10 seconds, immediately after first vasopressor dosage during standardised ALS-CPR procedures according to the International CPR Guidelines.

Group B (reference) Placebo, as a single IV bolus over 5-10 seconds, immediately after first vasopressor dosage during standardised ALS-CPR procedures according to the International CPR Guidelines.

ELIGIBILITY:
Patients, indicated for pre-hospital ALS-CPR procedures* must fulfil the following inclusion criteria:

* Age at least 18 years (known or estimated; no upper limit)
* Out-of-hospital cardiac arrest of presumed cardiac origin (including recurrent cardiac arrest(s) after initial ROSC)
* Witnessed (by eye and/or ear) cardiac arrest
* BLS-CPR started within 10 min of onset (known or estimated time) and may be performed for up to 10 min, followed by ALS-CPR - or ALS-CPR started within 10 min of onset (known or estimated time)

Subjects who meet any of the following criteria will be excluded from randomisation into the study:

* In-hospital cardiac arrest
* Cardiac arrest of presumed non-cardiac origin (e.g., drug overdose, carbon monoxide poisoning, drowning, hypothermia, exsanguination, electrocution, asphyxia, hypoxia, trauma, cerebrovascular accident)
* Obvious significant internal bleeding
* Known neurological impairment
* Known coagulation disorder
* Known pregnancy
* Known current participation in any other clinical study
* Known hypersensitivity to study medication
* Institutionalised subjects (e.g., prisoner)
* Any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050
Dates: Start 2004-01; Primary Completion 2006-06; Study Completion 2006-06

PRIMARY OUTCOMES:
The primary endpoint of this study is the 30-day survival rate | 30 days
The co-primary endpoint of this study is hospital admission | 30 days

SECONDARY OUTCOMES:
Return of spontaneous circulation (ROSC) | 30 days
24-hr survival | 24 hours
Neurological and overall outcome at hospital discharge or at day 30, whichever came first | 30 days
Symptomatic intracranial haemorrhage (ICH) up to hospital discharge or day 30, whichever came first | 30 days
Major bleeds up to hospital discharge or day 30, whichever came first | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (68):
- Austria (4):
  - Univ.-Klinik f. Anaesthesie Graz, Graz
  - Univ.-Klinik f. Anaesthesie u. Intensivmedizin, Innsbruck
  - LKH Salzburg, St. Johanns-Spital, Salzburg
  - Univ.-Klinik f. Notfallmedizin, Vienna
- Belgium (10):
  - Algemeen Ziekenhuis Antwerpen / Campus Stuivenberg, Antwerp
  - AZ Sint-Jan AV, Bruges
  - CHU Saint-Pierre, Brussels
  - AZ VUB, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Groeningen, Kortrijk
  - CHU de Tivoli, La Louvière
  - Universitaire Ziekenhuizen Leuven, Leuven
  - CHR de la Citadelle, Liège
  - CHR de Namur, Namur
- France (11):
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - Hôpital Henri Mondor, Créteil
  - Hôpital André Mignot, Le Chesnay
  - Hôpital Régional et Universitaire, Lille
  - Hôpital Marc Jacquet, Melun
  - Hôpital Lapeyronie, Montpellier
  - Hôpital Necker, Paris
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Purpan, Toulouse
  - Hôpital Pierre Bazin, Voiron
- Germany (17):
  - Universitätsklinikum Benjamin Franklin, Berlin
  - Humboldt-Klinikum, Berlin
  - DRK Kliniken Westend, Berlin
  - Städtische Kliniken Bielefeld gem. GmbH, Bielefeld
  - Klinikum der Ruhr-Universität Bochum, Bochum
  - Knappschaftskrankenhaus Dortmund, Dortmund
  - Chirurgische Universität Freiburg, Freiburg/Breisgau
  - Georg-August Universität Göttingen, Göttingen
  - Martin-Luther-Universität Halle, Halle
  - Universität Heidelberg, Heidelberg
  - Friedrich-Schiller Universität Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Berufsfeuerwehr Kiel, Kiel
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum rechts der Isar, München
  - Klinikum Saarbrücken gGmbH, Saarbrücken
  - Universitätsklinikum Ulm, Ulm
- Italy (6):
  - A. O. Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale S. Anna, Como
  - A. O. Universitaria S. Martino, Genova
  - A. O. San Gerardo di Monza, Monza
  - Policlinico S. Matteo, Pavia
  - Osp. di Circolo Fondazione Macchi, Varese
- Norway (4):
  - ICU, Haukeland Universitetssykehus, Bergen
  - ICU, Sykehuset Østfold Fredrikstad, Fredrikstad
  - Akuttklinikken / NLA, Sentralsjukehuset i Rogaland, Stavanger
  - Pre Hospital Klinikk, Sykehuset i Vestfold Tønsberg, Tønsberg
- Spain (10):
  - Hospital de Torrecárdenas / ICU, Almería
  - Hospital Clínico Provincial de BCN / Cardiology Service, Barcelona
  - Hospital Universitario Reina Sofía / ICU, Córdoba
  - Vírgen de las Nieves. Critical Care-Emergency Room, Granada
  - Hospital de Jerez de la Frontera / ICU, Jerez de la Frontera
  - Hospital Clínico San Carlos / Hemodynamics, Madrid
  - Hospital Clínico Universitario Vírgen de la Victoria / ICU, Málaga
  - Boehringer Ingelheim Investigational Site, Seville
  - Complejo Hospitalario Universitario de Vigo / Cardiology, Vigo
  - Hospital Clinico Univ. Lozano Blesa, Zaragoza
- Sweden (4):
  - Anestesikliniken, Gävle
  - Hjärt/Kärlforskn.enheten, Sahlgrenska Univ.sjh. Göteborg, Gothenburg
  - Universitetssjukhuset, Örebro
  - Södersjukhuset, Stockholm
- Switzerland (2):
  - Centre interdisciplinaire des urgences (CIU), CHUV BH 06-429, Lausanne
  - Boehringer Ingelheim Investigational Site, Lugano

REFERENCES:
- [Derived] Bottiger BW, Arntz HR, Chamberlain DA, Bluhmki E, Belmans A, Danays T, Carli PA, Adgey JA, Bode C, Wenzel V; TROICA Trial Investigators; European Resuscitation Council Study Group. Thrombolysis during resuscitation for out-of-hospital cardiac arrest. N Engl J Med. 2008 Dec 18;359(25):2651-62. doi: 10.1056/NEJMoa070570. PMID 19092151